CLINICAL TRIAL: NCT00473252
Title: Surveillance of Fungal Infections During Construction Activity
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Andreas Pasch, Department of Nephrology and Hypertension, Inselspital, University Hospital Bern
Other Study IDs: BE003
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Aspergillosis
Keywords: aspergillus infections; immunosuppression; kidney transplantation; hemodialysis; galactomannan test; fine dust; construction activity; airborne aspergillus spores
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis patients
- Renal transplant patients

SUMMARY:
Fungal infections in immunocompromised patients occuring during construction activities in hospitals have repeatedly been reported.

However, the question of a causal relation between construction activities and infections has never been addressed systematically and prospectively.

To answer this question, we will monitor our immunosuppressed patients' health status, as well as fine dust and aspergillus spore contents in the air during a three year construction activity period in our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation
* Chronic hemodialysis treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prevalent hemodialysis patients and incident renal transplant recipients in the Department of Nephrology and Hypertension, University Hospital Bern, Switzerland
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pasch, MD, Study Director — University of Bern
Locations (1):
- Dept. Nephrology & Hypertension, Univ. Hospital Bern, Bern, Canton of Bern, Switzerland